CLINICAL TRIAL: NCT04953988
Title: Technology and System for Minimally Invasive TKA Surgery Robot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M2021188
Record Dates: First submitted 2021-06-24; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Osteoarthritis, Knee
Keywords: KOA; TKA; robotic surgery
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Robotic surgery group (Experimental)
  Interventions: Procedure: Robotic TKA
- Manual operation group (Active Comparator)
  Interventions: Procedure: Manual operation

INTERVENTIONS:
Procedure: Robotic TKA — Robotic TKA
  Arms: Robotic surgery group
Procedure: Manual operation — Manual operation
  Arms: Manual operation group

SUMMARY:
Developed a robot for minimally invasive TKA surgery and prepare for the subsequent CFDA application of the minimally invasive total knee replacement robot system.

DETAILED DESCRIPTION:
1. For the current minimally invasive total knee arthroplasty, due to the limitation of the surgical field of view and the scope of operation, and the error of the intraoperative osteotomy saw, it can cause intraoperative damage to ligaments, nerves and blood vessels, postoperative lower limb force lines and prosthesis position Poor, abnormal movement and force of the patellofemoral joint and tibiofemoral joint after surgery can easily lead to clinical symptoms such as rapid wear of the prosthesis, short service life, postoperative knee pain, and even possible problems with surgical failure and revision. Developed a robot for minimally invasive total knee replacement surgery. Minimally invasive total knee arthroplasty is performed by surgical robot and manual operation. According to intraoperative and postoperative imaging observations, the position of the prosthesis, and the evaluation of soft tissue balance during and after the operation, the two methods are compared with the surgical robot and manual operation. Kind of surgery.
2. To prepare for the subsequent CFDA application of the minimally invasive total knee replacement robot system.

ELIGIBILITY:
Inclusion Criteria:

1. No surgery on the knee joint.
2. Age>55

Exclusion Criteria:

1. Knee surgery history.
2. Severe knee joint deformity (valgus greater than 15° or valgus greater than 20°) or knee joint instability.
3. Severe flexion contracture deformity.
4. Revision and replacement surgery for knee joints.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Full-length radiography of both lower limbs | Before and two days after the operation
  Measurement of lower limb force line and prosthesis position through full-length radiography of both lower limbs
Conventional anteroposterior radiograph of Both Lower Extremities | Before and two days after the operation
  Measurement of lower limb force line and prosthesis position through conventional anteroposterior radiograph of Both Lower Extremities
computed tomography | Before and two days after the operation
  Measurement of lower limb force line and prosthesis position through computed tomography
Magnetic Resonance Imaging | Before and two days after the operation
  Measurement of lower limb force line and prosthesis position through Magnetic Resonance Imaging
Range of motion | Before and two days after the operation
  Knee joint range of motion. Normal flexion 150°, extension 0°
Operation time | During the operation
  The time from the start of the skin incision to the completion of the skin suture